CLINICAL TRIAL: NCT00739531
Title: Measuring the Fractional Concentration of Exhaled Nitric Oxide (eNO) Using the Apieron INSIGHT System and the Aerocrine NIOX System
Brief Title: Measuring Exhaled Nitric Oxide (eNO) Using the Apieron INSIGHT System and the Aerocrine NIOX System
Status: Completed | Type: Observational
Sponsor: Apieron (Industry)
Responsible Party: Nina Peled, VP of Regulatory and Clinical Affairs, Apieron
Other Study IDs: CP00014
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Asthma
Keywords: Asthma; nitric oxide; eNO; FENO; Apieron INSIGHT; Aerocrine NIOX
MeSH Terms: conditions — Asthma | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthmatics: Subjects with asthma
  Interventions: Device: Exhaled nitric oxide (eNO)

INTERVENTIONS:
Device: Exhaled nitric oxide (eNO) — Subjects will perform a controlled breath maneuver using both the Apieron and NIOX devices. The devices will measure nitric oxide in the subjects' exhaled breath.

SUMMARY:
Collection of quantitative data to demonstrate the accuracy (bias) and precision (repeatability) of the Apieron INSIGHT(tm) eNO Breath System as compared to the FDA cleared NIOX eNO Breath System when testing is performed by asthma patients.

DETAILED DESCRIPTION:
A non-randomized, prospective study of up to 150 subjects with asthma. Patients will perform eNO testing with the Apieron INSIGHT(tm) eNO system and the NIOX eNO system at the physician's office/clinic after a short demonstration and training by a healthcare professional trained in the use of the devices. Exhaled NO testing involves inhaling to lung capacity, and then performing a controlled exhalation into a mouthpiece connected to each of the Apieron INSIGHT(tm) and NIOX systems. Patients will perform an eNO measurement with the Apieron INSIGHT(tm) system and with the FDA cleared NIOX system for the accuracy portion of the study. Patients will perform 2 sequential eNO measurements on each system for the precision part of the study. Subjects that measure eNO values over 100 ppb will be asked to repeat 2 sequential eNO measurements on each system.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 or older
* Pre-existing diagnosis of asthma
* Non-smoker

Exclusion Criteria:

* Chronic inflammatory lung disease other than asthma
* Medical conditions that preclude hand-eye coordination

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 150 asthma patients recruited from the site center's population of patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
eNO using Apieron INSIGHT(tm) System and Aerocrine NIOX at 50 ml/s | Single point in time

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Asthma- Allergy Clinic& Research Center, Shreveport, Louisiana
  - Allergy, Asthma & Dermatology Research Center, LLC, Lake Oswego, Oregon